CLINICAL TRIAL: NCT00857051
Title: Postpartum Support: Can we Facilitate the Transition to Motherhood?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Hibah Osman, MD, MPH, American University of Beirut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FM.HO.04
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-03

CONDITIONS: Stress
Keywords: Stress
MeSH Terms: interventions — Motion Pictures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): A 22 minute DVD that discusses common stressor in the early postpartum.
  Interventions: Other: Film
- 2 (Experimental): A 24 hour hotline available for the first 3 months postpartum.
  Interventions: Other: Hotline Service
- 3 (Experimental): Both the film and the hotline will be given to this arm.
  Interventions: Other: Hotline Service; Other: Film
- 4 (No Intervention): A CD of children's music will be given to mothers in this arm.

INTERVENTIONS:
Other: Hotline Service — A 24 hour hotline to answer questions about baby care or mother self-care. Hotline will be answered by a midwife and answers will be based on algorithms.
  Arms: 2; 3
Other: Film — A DVD addressing common stressors in the early postpartum.
  Arms: 1; 3

SUMMARY:
We are conducting a study to look interventions that may reduce stress in the postpartum period for first- time mothers. One of these interventions is an educational film that describes the common stressors that first-time parents go through in the early postpartum period. The other is a hotline service that women can call at anytime during the first 3 months postpartum to ask about problems she or the baby may be experiencing.

DETAILED DESCRIPTION:
The postpartum period is a very stressful experience for most mothers. It is generally accepted that women are physically and psychologically stressed during the postpartum. After delivery a woman may have worries about the health of her baby and her own health, as well as the changes in her body, their impact on her sexual life and her relationship with her husband. In addition, she may have financial concerns, concerns about breastfeeding, and be worried about bonding with her baby.

First-time mothers also have to adapt to their new role as mothers and may be worried about their abilities to take care of the baby. This may cause first-time mothers to develop postpartum depression and other emotional problems. First-time mothers can feel overwhelmed, exhausted, and isolated in their new roles.

We are conducting a study to look interventions that may reduce stress in the postpartum period for first- time mothers. One of these interventions is an educational film that describes the common stressors that first-time parents go through in the early postpartum period. The other is a hotline service that women can call at anytime during the first 3 months postpartum to ask about problems she or the baby may be experiencing. The hotline will be answered by a trained midwife.

Women will be recruited from all hospitals in Beirut after delivery and before they leave the hospital. If they agree to participate in the study, they will be randomly assigned to receive the film, the hotline service, both the film and the hotline service, or a CD containing children's songs. Women will be visited at home at 2 - 3 months after delivery by a researcher to complete questionnaires designed to measure stress, depression and anxiety in the postpartum.

Participants will not receive any financial compensation for participating in the study. Although women may benefit from the interventions, we will not know that until we complete the study. However, participation in this study may benefit mothers in the future if we find that the hotline or educational video are useful. There are no risks associated with participation in this study.

Confidentiality of the collected information will be ensured. All information collected will be used for research purposes and will be kept anonymous.

ELIGIBILITY:
Inclusion Criteria:

* Healthy first-time mothers with singleton baby delivered at term with no complications.

Exclusion Criteria:

* Mothers with chronic health problems,
* Pregnancy complications, OR
* Infants with congenital problems or conditions requiring admission to the intensive care nursery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 552 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Stress as measure by the Cohen Perceived Stress Scale (PSS-10) | 2 - 3 months

SECONDARY OUTCOMES:
Depression | 2 - 3 months
Anxiety | 2 - 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hibah Osman, MD, MPH, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon

REFERENCES:
- [Derived] Osman H, Saliba M, Chaaya M, Naasan G. Interventions to reduce postpartum stress in first-time mothers: a randomized-controlled trial. BMC Womens Health. 2014 Oct 15;14:125. doi: 10.1186/1472-6874-14-125. PMID 25315167
- [Derived] Hamade H, Chaaya M, Saliba M, Chaaban R, Osman H. Determinants of exclusive breastfeeding in an urban population of primiparas in Lebanon: a cross-sectional study. BMC Public Health. 2013 Jul 31;13:702. doi: 10.1186/1471-2458-13-702. PMID 23902627